CLINICAL TRIAL: NCT06365190
Title: Effects of a Periodic Repetitive Transcranial Magenetic Stimulation in Parkinson Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-PD-rTMS
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Transcranial Magnetic Stimulation; Parkinson's Disease
Keywords: Transcranial Magnetic Stimulation; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS group (Experimental): On the basis of drug treatment, a course of TBS treatment is performed every eight weeks.
  Interventions: Other: transcranial magnetic stimulation
- Drug group (Other): Take antiparkinsonian medications regularly, with follow-up every 8 weeks including medication guidance and symptom assessment
  Interventions: Drug: Pharmacotherapy（antiparkinsonian drugs）

INTERVENTIONS:
Other: transcranial magnetic stimulation — During treatment, the patient underwent cTBS targeting the left SMA for 14 consecutive days. Each treatment day comprised three rounds of cTBS, with a 15-minute interval between each. A single cTBS session involved trains of three pulses at 50 Hz, repeated every 200 ms (5 Hz), until reaching a total of 600 pulses, lasting 40s. Stimulation intensity remained at 80% of resting motor threshold. In total, patients received 25,200 pulses throughout the treatment period.
  Arms: cTBS group
Drug: Pharmacotherapy（antiparkinsonian drugs） — Anti-Parkinson's disease drugs include compound levodopa, dopamine receptor agonists, monoamine oxidase type B inhibitors, catechol-O-methyl transferase inhibitors, etc. Take dopaminergic agents regularly, with follow-up every 8 weeks including medication guidance and symptom assessment
  Arms: Drug group

SUMMARY:
Previous studies have shown that repetitive transcranial magnetic stimulation(rTMS) can improve clinical symptoms of Parkinson's disease(PD). Continuous theta-burst stimulation(cTBS) is a novel rTMS protocol that produces physiological effects b acting on neurons in the brain, which can decrease the excitability of motor system. This study aims to explore the long-term effects of cTBS on improvement of movement symptoms in patients with PD.

DETAILED DESCRIPTION:
This was a open-label clinical trial to assess the Effects of a Periodic Repetitive Transcranial Magenetic Stimulation in Parkinson Disease.

Participants were randomly assigned to the cTBS group and the control group on a 1:1 basis using age as a stratification factor. In the cTBS group, after baseline assessment, participants received cTBS treatment on the left supplementary motor area(SMA) for 14 days, and symptoms were assessed on the second day after treatment. Ten weeks after completion of assessment, a second cTBS session was performed, with all patients taking stable doses of antiparkinsonian medications. The control group only received drug intervention, and symptom assessment was conducted at weeks 13, 23 , 33 , and 43. To rule out the influence of medication on symptom assessment, all patients stopped taking medication for at least 12 hours before assessment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Chinese diagnostic criteria for Parkinson's disease (2016 version);
* Age ≥ 40 years old;
* Stable use of medication for at least 2 weeks;
* MMSE score ≧ 24 points;
* Those who can cooperate to complete the experiment; (6) Those who have not received rTMS treatment in the past.

Exclusion Criteria:

* History or clinical symptoms of other serious mental illnesses (such as major depression, psychosis, or obsessive-compulsive disorder);
* Severe organic brain defects on T1 or T2 images;
* History or unknown epilepsy Cause of loss of consciousness;
* Head injury, stroke or other neurological disease;
* Immovable metal objects on or around the head;
* History of drug abuse within the past 6 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale III scores | baseline; week 3; week 13;week 23;week 33
  This is an very common clinical motor estimating scale with 14 items and 108' in total. Higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
Hoehn-Yahr(H-Y) stage | baseline; week 3; week 13;week 23;week 33
  It ranges from 1 to 5, and is evaluated based on the range of symptoms involved and whether balance is impaired in PD patients. The higher the score, the more severe the severity.
Levodopa equivalent dose | baseline; week 3; week 13;week 23;week 33
  Different antiparkinsonian drugs converted to equivalent amounts of levodopa.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No